CLINICAL TRIAL: NCT06815614
Title: A Photoplethysmography-Based Continuous Automated Non-Invasive Sphygmomanometer: Performance Evaluation in Stability and Blood Pressure Change Tracking
Brief Title: This Study Aims to Assess the Performances of Optical Blood Pressure Monitoring Device, tBPC Product With Reference to ISO 81060-3:2022
Status: Completed | Type: Observational
Sponsor: Taiwan Biophotonic Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: tBPC-BP-202309072DS
Record Dates: First submitted 2025-01-12; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Blood Pressure; Blood Pressure Variability
Keywords: ISO 81060-3:2022; Photoplethysmography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: A Photoplethysmography-Based Continuous Automated Non-Invasive Sphygmomanometer — The investigation medical device under evaluation is oCareTM BP 100, a non-invasive continuous blood pressure monitoring system developed by Taiwan Biophotonic Co. (tBPC). The main function is to use a fingerclip sensor to receive PPG signals and collect continuous blood pressure values and uninterruptedly within the initialization time. In this study, according to the latest released ISO 81060-3:2022 standard requirements, non-invasive blood pressure measurement by cuff at the start and the end time points will be used as oCareTM BP 100 start-to-end blood pressure calibration. The A-line invasive arterial catheter blood pressure measurement will be used as a reference invasive BPM equipment. The purpose of the study is to confirm the stability of the investigational medical device under evaluation and its performance of blood pressure change tracking.

SUMMARY:
In this study, according to the latest released ISO 81060-3:2022 standard requirements, non-invasive blood pressure measurement by cuff at the start and the end time points will be used as oCareTM BP100 start-to-end blood pressure calibration. The invasive arterial catheter (A-line) blood pressure measurement will be used as a reference invasive blood pressure monitor (BPM) equipment. The purpose of the study is to evaluate the stability of the device under evaluation (DUE) and its performance in blood pressure change tracking.

DETAILED DESCRIPTION:
1. The primary goal (Stability Test): to validate the stability of the repeated measurements of DUE, and the corrected standard deviation of each analysis period shall not exceed 6 mmHg.
2. The secondary goal (Blood Pressure Change Tracking): to validate the consistency of DUE vs. the reference BPM equipment in blood pressure change tracking during the change evaluation interval.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be over 22 years old on the date of informed consent.
2. Subject who has undergone radial artery cannulation (A-line) (for medical purposes, specifically for arterial pressure monitoring.
3. Subject or his/her legal representative understand the written informed consent and willing to participate as evidenced by signing the informed consent.

Exclusion Criteria:

1. Pregnancy
2. Patients with an intra-aortic balloon pump
3. Patients with arm or finger injuries
4. Patients who have undergone vascular surgery for upper extremities or contraindications for local treatment upon upper extremities
5. Patients with A-line placement in the brachial artery
6. Participants are considered not suitable for inclusion after evaluation by the researchers (such as poor compliant mental status or health conditions, etc.)
7. Participants or his/her legal representative refuse to sign the informed consent form

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in the National Taiwan University Hospital Hsin-Chu Branch. A total of 30~40 patients are intended to be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Confirm the stability of the repeated measurements of SUT by calculating the corrected standard deviation of each analysis period | 4 hours
Confirm the consistency of SUT vs. the reference BPM equipment by calculating the blood pressure change during the change evaluation interval | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No